CLINICAL TRIAL: NCT03717740
Title: A Randomized Double-Blinded Placebo-Controlled Trial of Esomeprazole for the Prevention of Preeclampsia in Moderate- and High-Risk Women: The ESOPOP Trial
Brief Title: Esomeprazole for the Prevention of Preeclampsia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/291/9/18
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Pre-Eclampsia
Keywords: preeclampsia; esomeprazole; Soluble Fms Like Tyrosine Kinase -1
MeSH Terms: conditions — Pre-Eclampsia | interventions — Esomeprazole

STUDY DESIGN:
Intervention Model Description: The population of interest involves women attending the study hospital for antenatal care and delivery. The intervention involves randomization to oral esomeprazole tablets40 mg or identical placebo tablet from recruitment until delivery. Randomization is achieved using computational random allocation, and both participants and researchers will be blinded to the intervention given.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: both participants and researchers will be blinded to the intervention given.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esomeprazole (Experimental): Patients will take esomeprazole single dose of 40 mg orally once a day from 12+ and 17 weeks of pregnancy until 34 weeks of pregnancy,
  Interventions: Drug: Esomeprazole
- Placebo (Placebo Comparator): Patients will take Placebo Oral Tablet once a daily oral tablet from 12+ and 17 weeks of pregnancy until 34 weeks of pregnancy,
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — Patients will take esomeprazole single dose of 40 mg orally once a day from 12+ and 17 weeks of pregnancy until 34 weeks of pregnancy
  Other Names: Experimental
  Arms: Esomeprazole
Drug: Placebo — Patients will take an inert tablet similar in appearance, color, and consistency from 12+ and 17 weeks of pregnancy until 34 weeks of pregnancy
  Other Names: Placebo Comparator
  Arms: Placebo

SUMMARY:
Preeclampsia, one of the hypertensive disorders of pregnancy, remains a leading cause of maternal death worldwide, with the majority of deaths occurring in developing countries. Preeclampsia is a multi-organ syndrome of pregnancy that manifests after 20 weeks' gestation with new-onset hypertension alongside maternal end-organ dysfunction and/or fetal growth restriction. Importantly, preeclampsia poses serious health risks for the baby, implicated in 12% of cases of fetal growth restriction, and is a known antecedent in up to 19% of preterm births. There is currently no effective treatment for preeclampsia except delivery of the baby, and as such, it remains a significant burden of disease for both mothers and their babies worldwide. Screening for women at risk of preeclampsia is an important part of antenatal care. Once women are identified as high risk, they can be targeted for more intensive antenatal surveillance and prophylactic interventions. Most current strategies for risk assessment are based on obstetric and medical history and clinical examination. However, there is surprisingly little reliable evidence on the actual risk associated with individual factors and how they might interact. Risk factors with a particularly high association with preeclampsia (more than one in ten risks) include maternal diabetes, chronic hypertension, and renal disease. Thrombophilia and autoimmune disease have a strong association with severe early-onset preeclampsia. Obstetric factors associated with high risk are multiple pregnancies, history of preeclampsia in a previous pregnancy especially if severe or early onset, and a current hydropic pregnancy. Other factors linked with preeclampsia but associated with a somewhat lower risk include first pregnancies, age less than 20 or more than 35 years, a family history of preeclampsia, and obesity. Proton pump inhibitors such as esomeprazole have long-term safety data about the treatment of gastric reflux in pregnancy. In vitro studies show proton pump inhibitors decrease soluble fems like tyrosine kinase -1 (sFlt-1) and soluble endoglin and improve markers of endothelial dysfunction . while esomeprazole reduces blood pressure in a preeclampsia transgenic mouse model that overexpresses sFlt-1.

DETAILED DESCRIPTION:
This is a randomized double-blinded placebo-controlled intervention trial investigating preeclampsia, defined according to the National Institute of Clinical Excellence (NICE). The population of interest involves women attending the study hospital for antenatal care and delivery with a risk for developing preeclampsia. The intervention involves randomization to oral esomeprazole tablets40 mg or identical placebo tablet from recruitment until delivery. Randomization is achieved using computational random allocation, and both participants and researchers will be blinded to the intervention given. Calculation of the sample size considers that the incidence of preeclampsia is 10% in the population of interest. To detect a 50% reduction in incidence (with 80% power, two-sided p < 0.05), 450 women are required in each group with a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women presenting prior to 17+0 weeks' gestation.

  * Moderate to high risk of preeclampsia. One or more of the following: previous history of preeclampsia, antiphospholipid antibodies, pre-existing diabetes, pre-existing hypertension, pre-existing renal disease, autoimmune disease, nulliparity, family history of preeclampsia, elevated BMI > 25, and maternal age <20 or >35.
* Give written informed consent.

Exclusion Criteria:

* Multiple pregnancies.
* Current or previous esomeprazole ingestion within the last 6 weeks.
* Previous hypersensitivity reaction esomeprazole
* Contraindications to the use of a proton pump inhibitor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The population of interest involves women attending the study hospital for antenatal care and delivery
Enrollment: 1000 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With early onset Preeclampsia | 6 months
  The number of cases of preeclampsia that appear in both groups before 34 weeks of pregnancy.Blood pressure greater than 140/90 on 2 occasions 6 hrs apart and significant proteinuria (greater than 300 mg in 24 hrs) before 34 weeks gestation

SECONDARY OUTCOMES:
Prevention of preeclampsia between 37 and 41 | 6 months
  The number of cases of preeclampsia that appear in both groups between 37 and 41 weeks of pregnancy.
The number of cases of Fetal Growth Restriction | 6 months
  The number of cases of fetal growth restriction, defined as a fetal weight below the 10th percentile and an abnormal umbilical cord doppler that appear in both groups at any given time during pregnancy.
The number of cases of preterm birth | 6 months
  The number of cases delivered before complet 37 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No